CLINICAL TRIAL: NCT06403995
Title: Evidence-based Internet Cognitive-behavioral Therapy for Social Anxiety
Acronym: iCBT-SAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-4843
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Social Anxiety
Keywords: Anxiety; Social anxiety; Internet Cognitive behavioural therapy; Community-based primary health care; Quasi-experimental design; Canada
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Individuals with social anxiety will either: 1) self-refer to the adapted intervention (self-referral, undirected iCBT); 2) be recommended the adapted intervention by a registered health professional and will complete the program without guidance (recommended, undirected iCBT); or 3) be recommended the adapted intervention by a registered health professional, with low-intensity guidance throughout the program (recommended, directed iCBT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Self-referred, undirected iCBT (Experimental): These individuals will do the program, but will not receive follow-up contact during the program. In case of severe psychological distress (i.e. score ≥30 on Kessler's 10-item psychological distress scale (K10), participants will receive an automated email with a list of resources and emergency contact numbers.
  Interventions: Behavioral: Self-referred, undirected Internet-based cognitive behavioral therapy for social anxiety
- Recommended, undirected iCBT (Experimental): Participants will have received the recommendation from a healthcare professional (e.g., family physician, nurse or social worker, psychologist) to complete the adapted program without guidance. Clinicians will provide the name and email of the patients they are referring the program to without providing participants with in-program support but will consult the dashboard as they have clinical responsibility for the patient. In case of severe distress (i.e., K10 score ≥30), the referring healthcare professional will receive an automated email informing them to go to their dashboard to identify that patient. Participants will also receive an automated email with a list of resources and emergency contact numbers. To support the generalization of findings to the real-world (ecological validity), clinicians may follow-up with patients at their discretion.
  Interventions: Behavioral: Recommended, undirected Internet-based cognitive behavioral therapy for social anxiety
- Recommended, directed iCBT (Experimental): Participants will be recommended the intervention by a healthcare professional and be provided low-intensity guidance (e.g., email or brief phone contact [5 to 10 minutes] after Lesson 1 and 2, and then on an as-needed basis or patient request). Clinicians at the primary care sites participating in the study will be able to recommend the adapted program to their patients, will remain responsible for their patients and, will check their dashboard to see how their patients are progressing through the program. In the event of severe distress (i.e., K10 score ≥30) in a patient, the referring healthcare professional will receive an automated email informing them to go to their dashboard to identify that patient and assess the appropriate action to take. Participants will also receive an automated email with a list of resources and emergency contact numbers.
  Interventions: Behavioral: Recommended, directed Internet-based cognitive behavioral therapy for social anxiety

INTERVENTIONS:
Behavioral: Self-referred, undirected Internet-based cognitive behavioral therapy for social anxiety — The Shyness Program is presented in the form of illustrated stories of a working woman and young man with SAD and their health professional (a psychologist). The program comprises six online lessons that teach core cognitive and behavioral principles and skills, including psychoeducation about the symptoms and treatment of SAD (Lessons 1-2); graded exposure and behavioral experiments (Lesson 3); cognitive restructuring (Lessons 4-5); relapse prevention (Lesson 6). The program also includes lesson summaries, homework assignments, and regular scheduled emails to support program users in applying the CBT skills themselves (N. Titov, Andrews, Schwencke, et al., 2008). It is recommended that modules are completed every 1 to 2 weeks with the full program completed within 90 days (see https://thiswayup.org.au/courses/the-social-anxiety-course/).
  Arms: Self-referred, undirected iCBT
Behavioral: Recommended, undirected Internet-based cognitive behavioral therapy for social anxiety — The Shyness Program is presented in the form of illustrated stories of a working woman and young man with SAD and their health professional (a psychologist). The program comprises six online lessons that teach core cognitive and behavioral principles and skills, including psychoeducation about the symptoms and treatment of SAD (Lessons 1-2); graded exposure and behavioral experiments (Lesson 3); cognitive restructuring (Lessons 4-5); relapse prevention (Lesson 6). The program also includes lesson summaries, homework assignments, and regular scheduled emails to support program users in applying the CBT skills themselves (N. Titov, Andrews, Schwencke, et al., 2008). It is recommended that modules are completed every 1 to 2 weeks with the full program completed within 90 days (see https://thiswayup.org.au/courses/the-social-anxiety-course/).
  Arms: Recommended, undirected iCBT
Behavioral: Recommended, directed Internet-based cognitive behavioral therapy for social anxiety — The Shyness Program is presented in the form of illustrated stories of a working woman and young man with SAD and their health professional (a psychologist). The program comprises six online lessons that teach core cognitive and behavioral principles and skills, including psychoeducation about the symptoms and treatment of SAD (Lessons 1-2); graded exposure and behavioral experiments (Lesson 3); cognitive restructuring (Lessons 4-5); relapse prevention (Lesson 6). The program also includes lesson summaries, homework assignments, and regular scheduled emails to support program users in applying the CBT skills themselves (N. Titov, Andrews, Schwencke, et al., 2008). It is recommended that modules are completed every 1 to 2 weeks with the full program completed within 90 days (see https://thiswayup.org.au/courses/the-social-anxiety-course/).
  Arms: Recommended, directed iCBT

SUMMARY:
The objectives of the study are to 1) to translate and adapt iCBT Shyness Program to the Canadian context; 2) to examine the completion and effectiveness of the Canadian adapted, including the French translated and English iCBT Shyness Program, in improving SAD symptoms; 3) to explore barriers and facilitating factors to the program's implementation. The overall study design is a hybrid effectiveness-implementation study of a quasi-experimental parallel group trial reflecting real world pathways (recommended and self-referrals). The project will be conducted in two Canadian provinces: Quebec (Montérégie) and Ontario. Prior to implementing the iCBT Shyness Program, it will undergo an initial adaptation to the Canadian context and focus groups will be conducted with key actor groups to discuss the adaptations to the graphics, narration of the modules, and this to better reflect varying sociocultural context among Canadian French- and English-speaking populations. We will then evaluate the outcomes associated with the implementation of the program in a three-pathway parallel trial. As a last step to this trial, semi-structured interviews will be conducted with study participants and health care providers to explore facilitating factors and barriers to the implementation of the iCBT adapted program.

DETAILED DESCRIPTION:
Study rational Social anxiety disorder (SAD) is one of the most prevalent anxiety disorders, with lifetime and past-year prevalence estimates reaching 12% and 7% in Canada. In the absence of treatment SAD is a chronic disorder with significant impairment in functioning associated with reduced school performance, loss of productivity, and decreased quality of life. During COVID-19, studies highlight increased mental health needs, but barriers to mental health service access due inpart to limited resources available. Viable therapy options for the treatment of SAD include CBT being delivered virtually, with effectiveness being shown in youth and adults. The Clinical Research Unit for Anxiety and Depression (CRUfAD) in Australia has developed, implemented, and demonstrated the effectiveness of an innovative guided and unguided internet delivered cognitive-behavioural therapy (iCBT) program for social anxiety. To make available high-quality and real-time evidence in response to the current COVID-19 mental health crisis and crucially needed access to psychological services to meet population mental health needs including for high risk populations (including individuals with pre-existing psychiatric conditions, youth and young adults, self identifying as belonging to a visible minority group (including from linguistic minority groups), we propose to conduct a Canadian adaptation of Australia's Shyness Program and to examine the adapted program's effectiveness, and implementation in two Canadian provinces (Quebec and Ontario).

Objectives

1) to translate and adapt iCBT Shyness Program to the Canadian context; 2) to examine the completion and effectiveness of the Canadian-adapted, including the French translated and English iCBT Shyness Program, in improving SAD symptoms; 3) to explore barriers and facilitating factors to the program's implementation.

Methods

The overall study design is a hybrid effectiveness-implementation study of a quasi-experimental parallel group trial reflecting real world pathways (recommended and self-referrals). The project will be conducted in two Canadian provinces: Quebec (Montérégie) and Ontario.

To build on the current knowledge regarding the effectiveness of guided and unguided iCBT for SAD and inform on generalizability, we will evaluate the outcomes associated with the implementation of the program in a three-pathway parallel trial. The iCBT Shyness Program includes six online lessons based on CBT strategies with homework assignments to be completed within 90 days. The study will be carried out in Quebec and Ontario.

Phase 1:

Prior to implementing the iCBT Shyness Program, it will undergo an initial adaptation to the Canadian context. Focus groups in each province will be conducted with key actor groups (patients-partners, community leaders, service providers, i.e., consultant-partners to the research team) to discuss the adaptations to the graphics, narration of the modules, and this to better reflect varying sociocultural context (e.g., socioeconomically disadvantaged environment; cultural backgrounds) among Canadian French- and English-speaking populations.

Phase 2:

Then, individuals with social anxiety will either: 1) self-refer to the adapted intervention (self referral, undirected iCBT); 2) be recommended the adapted intervention by a registered health professional and will complete the program without guidance (recommended, undirected iCBT); or 3) be recommended the adapted intervention by a registered health professional, with low intensity guidance throughout the program (recommended, directed iCBT). The program will be implemented via the virtual clinic at Université de Sherbrooke (www.equilia.ca), as we have acquired and implemented a license for the virtual clinic in Canada. Data collection will be integrated into the virtual clinic web platform and the REDCap platform and carried out at baseline, at the beginning of each lesson, 12-week and 6-month follow-up. Individual-level outcomes measured will include anxiety and depressive symptoms, psychological distress, disability, health-related quality of life as well as health service utilization and satisfaction.

Phase 3:

As a last step to this trial, semi-structured interviews will be conducted with study participants and health care providers to explore facilitating factors and barriers to the implementation of the iCBT adapted program, and this to inform implementation strategies for wider use across Canada.

Anticipated results

This study will provide evidence on the effectiveness, barriers and facilitating factors to implementing a low-intensity iCBT in the Canadian context for SAD, which will bridge an important care gap for undeserved populations in Canada with SAD. Findings will inform the eventual scaling up of the program in community-based primary health care across Canada. This would improve equity of the health care system by helping a large number of Canadians including those from visible, socio-cultural, and linguistic minority groups timely access to mental health services post-pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years; and
* Speak and write in French or English; and
* Have access to the internet and a digital device; and
* Screen for social anxiety using the 17-item Social Phobia Inventory (SPIN) questionnaire (> 20).

Exclusion Criteria:

* Self-report severe symptoms of depressions (PHQ-9 score ≥ 23); or
* Thoughts they would be better off dead or hurting themselves on the 9th item of PHQ-9 in the past two weeks or thoughts or wishes to kill themselves on the 9th item of the Beck Depression Inventory-II; or
* A diagnosis of schizophrenia, bipolar disorder or problems related to active substance use or dependence; or
* Current use of benzodiazepines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change on the Social Phobia Inventory (SPIN) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Social Phobia Inventory (SPIN). The 17-item SPIN questionnaire will be used to assess social anxiety symptoms, which are rated on a 5-point scale from 0 (not at all) to 4 (extremely), with a possible score range from 0 to 68 (Connor et al., 2000). A cut-off > 20 has been shown to reflect a probable case of SAD (Davidson, 2020).

SECONDARY OUTCOMES:
Change on the World Health Organization Disability Assessment Schedule (WHODAS 2.0) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) (Andrews, Kemp, Sunderland, Von Korff, & Ustun, 2009). The 12-item schedule measures activity limitations in the past 30 days in 6 domains (possible score range 0 to 60), will also be used to assess disability.
Change in Health-related quality of life (HRQOL) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Health-related quality of life (HRQOL) will be ascertained with the four-dimension Assessment of Quality of Life (AQoL-4D) (Hawthorne G, Richardson J, Osborne R, 1999; Hawthorne G, Richarson J, Day NA, 2001) including 12 items on 4 dimensions: independent living, mental health, relationships, senses. Scoring will be based on available weights and utility scores range from 0 to 1.0 (AQol, 2014; Richardson et al., 2014).
Change on the Kessler Psychological Distress Scale (K10) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Kessler Psychological Distress Scale (K10) (Kessler et al., 2002). The 10-item scale assesses psychological distress on a 5-point scale with scores ranging from 10 to 50. Scores ≥30 correspond to severe distress and an alert is sent to the study team, the participant, and referring health professional.
Change in Patient Health Questionnaire-8 (PHQ-8) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Patient Health Questionnaire (PHQ-8). The 8-item questionnaire will be used to assess depressive symptoms. Symptoms are rated on a 0 (not at all) to 3 (nearly every day) point scale, with scores ranging from 0 to 24. A cut-off score ≥10 is used to identify a probable major depressive disorder (Kroenke et al., 2009).
Change in generalized anxiety disorder scale (GAD-7) | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Generalized Anxiety Scale (GAD-7). The 7-iem questionnaire will be used to assess generalized anxiety symptoms with scores ranging from 0 to 21. A cut-off score ≥10 is used to identify probable anxiety (Spitzer, Kroenke, Williams, & Löwe, 2006).
Past 3 and 6-month health and social service use | Baseline and 6-month post-treatment
  Past 3 and 6-month health and social service use (any emergency department visit, any hospitalisation, visit to a health professional, receipt of services from local community service centre, psychotropic drug use).
Self-reported satisfaction with iCBT program | 12-week post-treatment
  As in Williams et al., (2014) (Williams et al., 2014), self-reported satisfaction with the iCBT program will be assessed with a 5-point scale assessing how satisfied individuals were with the program: 1= very dissatisfied to 5=very satisfied; and how confident participants are in recommending the program to a family member/friend with social anxiety (1=not at all to 10= extremely confident).
Contacts with referring prescriber | 6-month post-treatment
  Number of contacts (e.g. consultations) with referring prescriber of the program

OTHER OUTCOMES:
Change in loneliness and social isolation | Baseline to post-treatment (12-week and 6-month follow-up post-treatment)
  Loneliness will be assessed using the 6-item Revised UCLA Loneliness Scale measured on a 4-level Likert scale (I often/sometimes/rarely/never feel this way) with a total score ranging from 0 to 24 (Wongpakaran N, Wongpakaran T, Pinyopornpanish M, Simcharoen S, Suradom C, Varnado P, Kuntawong P, 2020).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CISSS de la Montérégie-Centre, Greenfield Park, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
The authors are not legally authorised to share or publicly publish participants' data. Participants were not requested to give informed consent for public data sharing. Requests for access to the data should be addressed to the Ethics Committee Board of the Centre Intégré Universitaire de Santé et Services Sociaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke.

REFERENCES:
- [Derived] Vasiliadis HM, Roberge P, Spagnolo J, Lamoureux-Lamarche C, Chapdelaine A, Brodeur M, Grenier J, Mahoney A, Koszycki D, Chomienne MH, Drapeau M, Labelle R, Provencher MD, Ishimo MC, Naslund JA, Lesage A. A digital iCBT intervention for social anxiety disorder in Quebec and Ontario: protocol for a multi-phase effectiveness-implementation study. BMC Psychiatry. 2024 Oct 8;24(1):662. doi: 10.1186/s12888-024-06082-7. PMID 39379845